CLINICAL TRIAL: NCT04360161
Title: Morphology of Schlemm's Canal and Crystalline Lens in Different Age: a Swept-source Optical Coherence Tomography Study
Brief Title: Observing the Morphology of Schlemm's Canal and Crystalline Lens in Different Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Director of Cataract Department, Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TM/SC/Lens-LZL
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Schlemm's Canal Occlusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy participants (Experimental): Swept-source optical coherence tomography A device testing TM/SC and Lens morphology
  Interventions: Device: swept-source optical coherence tomography

INTERVENTIONS:
Device: swept-source optical coherence tomography — Aswe pt-source OCT (CASIA SS-1000; Tomey Corporation, Nagoya, Japan), which is specifically designed for anterior segment imaging using a 1310 nm wavelength with a scan speed of 30,000 A-scans per second and an axial resolution of <10 μm.

SUMMARY:
The aim of this study is to quantify and observe the morphology of trabecular meshwork (TM), Schlemm's canal (SC), ciliary body and crystalline lens before and after cycloplegia in patients with different ages using swept-source optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients who can cooperated with the swept-source OCT measurements

Exclusion Criteria:

* history of ocular disease
* presence of central nervous system or systemic disease

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
area of Schlemm's canal and trabecular meshwork | up to 6 months
  The area of Schlemm's canal and trabecular meshwork was manually measured and the relationship between the parameters and age was analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Yune Zhao, Study Director — Eye Hospital of Wenzhou Medical University
Locations (1):
- Eye Hospital of WMU, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No